CLINICAL TRIAL: NCT00982267
Title: A Phase I Dose Escalating Study Of SU014813 In Patients With Solid Tumors Not Amenable To Conventional Therapy
Brief Title: A Trial Of SU14813 In Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTKD-7840-002; A6191002
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Neoplasms; Solid Tumors
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SU014813 (Experimental)
  Interventions: Drug: SU014813

INTERVENTIONS:
Drug: SU014813 — Escalating doses of SU014813 from 50 to 250mg/day . Capsules administered daily either as continuous dosing or in cycles of 4 weeks on 1 week off

SUMMARY:
The purpose of this study is to define the Maximum tolerated dose of SU14813 when administered as single agent in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically proven advanced solid malignancy for which no recognized therapy was available or for which standard therapy had failed
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Serum albumin ≥3.0 g/dL and adequate haemopoietic, renal and liver function

Exclusion Criteria:

* Chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy or an investigational agent within 4 weeks before the start of study treatment
* Subjects had to have recovered from all prior treatment toxicities, except alopecia, and from any major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-12; Primary Completion 2008-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 18-Nov-2008

SECONDARY OUTCOMES:
Determine the recommended Phase 2 dose (RP2D) | 18-Nov-2008
Preliminary information on SU014813 anti-tumor effect; | 18-Nov-2008
Plasma pharmacokinetics | 18-Nov-2008
Plasma targets such as vascular endothelial growth factor (VEGF), soluble VEGF-R2 and soluble KITa | 18-Nov-2008

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Hamburg, Germany
- Pfizer Investigational Site, Amsterdam, Netherlands

REFERENCES:
- [Derived] Fiedler W, Giaccone G, Lasch P, van der Horst I, Brega N, Courtney R, Abbattista A, Shalinsky DR, Bokemeyer C, Boven E. Phase I trial of SU14813 in patients with advanced solid malignancies. Ann Oncol. 2011 Jan;22(1):195-201. doi: 10.1093/annonc/mdq313. Epub 2010 Jul 6. PMID 20605934
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=RTKD-7840-002&StudyName=A%20Trial%20Of%20SU14813%20In%20Patients%20With%20Advanced%20Solid%20Malignancies